CLINICAL TRIAL: NCT00004334
Title: Study of Depression, Peptides, and Steroids in Cushing's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Other Study IDs: NCRR-M01RR00042-1781; UMMC-701
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's syndrome; endocrine disorders; rare disease
MeSH Terms: conditions — Cushing Syndrome; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Study the relationship between dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis and disorders of mood, vegetative function, and cognition in patients with Cushing's disease.

II. Identify subgroups of patients with Cushing's disease who differ in the presence and severity of the depressive syndrome, and uncover HPA axis dysregulation differences among them using corticotropin-releasing hormone, metyrapone, and dexamethasone challenge testing.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: All patients receive a psychiatric evaluation at baseline, as well as assessments of plasma adrenocorticotropin, beta lipotropin, beta endorphin, and cortisol, and urinary cortisol. Peptide and steroid assays are performed, alone and in response to corticotropin-releasing hormone, metyrapone, and dexamethasone. Patients are given sleep electroencephalograms at baseline and 1 year following treatment.

A weight maintenance diet is prescribed for all patients.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Patients aged 20 to 60 with spontaneous active Cushing's syndrome
* At least 2 weeks since medication with psychoactive effects or influence on cortisol metabolism by hepatic hydroxylating enzyme induction
* Antihypertensives allowed for severe hypertension
* No barbiturates
* No phenytoin

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8
Dates: Start 1994-07

CONTACTS AND LOCATIONS:
Overall Officials: Monica N. Starkman, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States